CLINICAL TRIAL: NCT03479606
Title: A Randomized Controlled Trial of an Online Emotion Regulation Intervention Following TBI
Brief Title: Online Emotion Regulation Group Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kristen Dams-O'Connor, Professor, Rehabilitation Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GCO 17-0988; IRB-17-02795 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2018-03-12; First posted 2018-03-27 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Traumatic Brain Injury; Executive Dysfunction; Emotion Dysfunction; Emotion Dysregulation
Keywords: Traumatic Brain Injury; TBI; Executive Dysfunction; Emotional Regulation; Emotional Dysfunction; Problem Solving; Self-regulation; Cognitive Rehabilitation; Metacognitive Strategies; Cognitive-behavioral therapy; Online Therapy; GroupTherapy; Group videoconference; Telehealth; Telerehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic; Emotional Regulation; Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Participants will receive 24 online emotional regulation skills-training sessions twice weekly and will complete online questionnaires sent every four weeks throughout baseline, the 12-week intervention, and 12-week follow-up.
  Interventions: Behavioral: Online Emotion Regulation Skills-training
- Waitlist Intervention (Active Comparator): After a 12-week wait-period without any intervention, participants will receive 24 online emotion regulation skills-training sessions. Every four weeks, participants will complete online questionnaires every throughout baseline, 12-week wait-period, 12-week intervention, and 12-week follow-up.
  Interventions: Behavioral: Online Emotion Regulation Skills-training

INTERVENTIONS:
Behavioral: Online Emotion Regulation Skills-training — Emotion Regulation Training (EmReg) is a cognitive-behavioral approach which aims to increase awareness, and self-monitoring of affective states to improve self-regulation. The intervention is divided into two phases: knowledge provision and practice facilitation. During the knowledge provision phase participants are introduced to the objectives and the main concepts of the intervention, to increase their familiarity with the terminology, and to the emotion regulation skills they acquire during the practice facilitation phase. During the practice facilitation phase participants receive training in emotion regulation skills, which they practice in-session with the guidance of the therapist and feedback from the group, as well as out-of-session as homework assignments.
  Other Names: Emotion Regulation Training (EmReg)

SUMMARY:
This study will examine the efficacy of an emotion regulation intervention delivered online to individuals with traumatic brain injury (TBI) with deficits in emotion regulation. 104 subjects will be enrolled and will receive 24, 60-minute emotion regulation skills-training sessions twice a week for 12 weeks, delivered online in a group video-conference with 3-5 other participants. Participants will be asked to complete online surveys, lasting approximately 40-50 minutes, every four weeks during the intervention and the 12-week follow-up phase. Attendance and compliance will be tracked, and outcomes will be monitored using online data collection methods.

DETAILED DESCRIPTION:
This study will assess the efficacy of an emotion regulation skills-training intervention (Online EmReg) provided online to individuals with TBI with emotion regulation difficulties. Specifically, this study seeks to accomplish three aims: 1) Evaluate the efficacy of the Online EmReg intervention immediately post-intervention and at a 12-week follow-up assessment; 2) Identify factors that optimize the effectiveness of the Online EmReg intervention; 3) Explore the impact of Online EmReg on positive and negative affect, life satisfaction, and executive functioning. The study design is a randomized control trial with a waitlist control group whereby the participants in the control group undergo the training after a 12 week waiting period. 104 subjects with TBI and self-reported deficits in emotion regulation will be enrolled.

The intervention protocol calls for 24, 60-minute emotion regulation sessions twice a week for 12 weeks, delivered online via Zoom by post-doctoral level therapists with specialty training in rehabilitation neuropsychology. Study participation will last approximately 28 weeks for participants in the immediate intervention arm (4 weeks preparation, 12 weeks intervention, 12 weeks follow-up) and 40 weeks for participants in the waitlist arm (4 weeks preparation, 12 weeks waitlist, 12 weeks intervention, and 12 weeks follow-up). Core assessments will be conducted at each major time point: T1 (baseline), T2 (immediate intervention end/waitlist baseline), T3 (immediate intervention follow-up/end of waitlist intervention), and T4 (waitlist follow-up). A subset of the measures will be administered every 4 weeks between each major time point for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* medically documented mild to severe TBI
* at least 6 months post-injury
* deficits in emotional regulation (ER), operationalized as a score of 0.5 standard deviations above published means on the Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004)
* English speaking
* adequate communication skills, assessed by the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC)
* access to and ability to use a device that supports GoToMeeting/Zoom, the videoconference software
* active email address
* access to the Internet with adequate broadband
* Lives in the following states for the duration of the 12-week intervention: New York, California, Maryland, North Carolina, Georgia, Missouri, Arizona, New Jersey, Colorado, Florida, or Washington DC

Exclusion Criteria:

* current alcohol or substance abuse
* current psychotic disorder, mood disorder with psychotic features or current suicidality, assessed by the Mini International Neuropsychiatric Interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | Every 4 weeks for 28 or 40 weeks
  36-item self-report questionnaire that focuses on emotional awareness, acceptance, ability to control impulsivity, and flexible use of strategies.

SECONDARY OUTCOMES:
Positive Affect Negative Affect Schedule (PANAS) | Every 4 weeks for 28 or 40 weeks
  A 20-item measure with two independent scales, positive affect and negative affect.
Satisfaction with Life Scale (SWLS) | Every 4 weeks for 28 or 40 weeks
  A 5-item measure of satisfaction with life globally.
Problem Solving Inventory (PSI) | Every 4 weeks for 28 or 40 weeks
  A 35-item self-report measure assessing problem solving behavior and attitudes, the PSI yields 3 subscales: Approach/Avoidance Style, Problem Solving Confidence, and Presence of Personal Control.
Dysexecutive Functioning Questionnaire (DEX) | Every 4 weeks for 28 or 40 weeks
  A 20-item sensitive and ecologically valid questionnaire assessing everyday problems.
Transition Ratings (TR) | End of intervention (at 16 or 28 weeks) and follow-up at 12-weeks post intervention
  These ratings are used to assess change on problems that are intervention targets, from the participant's point of view, by reporting how much better/worse the problem seems to be since the onset of the intervention.
Progress Toward Goals (PTG) | Every 4 weeks for 28 weeks
  During the first 2 sessions, participants will be asked to set three to five personal goals related to emotional regulation and its impact on their daily lives, and then asked to rate their progress towards these goals on a 7-point Likert scale.
Skill Acquisition Quiz (SAQ) | End of intervention (at 16 or 28 weeks) and follow-up at 12-weeks post intervention
  A 20-question content-based quiz developed to assess how well participants learn and retain EmReg concepts and strategies by intervention end.

OTHER OUTCOMES:
Access to Care Questionnaire (ACQ) | Baseline
  A brief questionnaire to assess participants' access to rehabilitation services using modified items borrowed from national health surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kajankova, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Kristen Dams-O'Connor, PhD, Study Director — Icahn School of Medicine at Mount Sinai; Theodore Tsaousides, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Brain Injury Research Center at Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No